CLINICAL TRIAL: NCT04454060
Title: Study on the Development of Arthroscopic Treatment of Refractory Tennis Elbow
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018063
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Tennis Elbow
Keywords: Qualitative; Quantitative; Tennis Elbow; Arthroscopy; Surgical Techniques
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extracapsular method group: consecutive 43 patients who received extracapsular method treatment for refractory tennis elbow
  Interventions: Procedure: Extracapsular arthroscopy

INTERVENTIONS:
Procedure: Extracapsular arthroscopy — Extracapsular arthroscopy method was used to treat refractory tennis elbow

SUMMARY:
The aim of this study was to investigate the exploration history, key theories, methods, and techniques involved in the evolution from the intracapsular method to the extracapsular method for arthroscopic treatment of tennis elbow, and explore the effectiveness and safety of extracapsular method on the basis of retrospective analysis of 43 cases.

DETAILED DESCRIPTION:
Background: Arthroscopic surgery is widely used in the treatment of refractory tennis elbow due to its advantages of minimally invasive, safe and direct vision. Intra-capsular arthroscopy(intracapsular method), which is performed via natural cavity, is the mainstream arthroscopic procedure. However, intracapsular method requires the damage of joint capsule and may cause intraoperative neurovascular injury and other complications. In view of the defects of intracapsular method, the surgical scheme of the extracapsular arthroscopy (referred to as "extracapsular method") has emerged. The aim of this study was to investigate the exploration history, key theories, methods, and techniques involved in the evolution from the intracapsular method to the extracapsular method for arthroscopic treatment of tennis elbow, and explore the effectiveness and safety of extracapsular method.

Methods: Qualitative data were collected via focus group interview. 7 surgeons who were selected through purposive sampling discussed on the theories, methods, and technical specifications of the transition from intracapsular method to extracapsular method. Qualitative data were analysed using NVivo11. Quantitative data of consecutive 43 patients were analysed to evaluate the effectiveness and safety of the extracapsular method. Descriptive analysis was conducted to analyse the demographic characteristics and clinical outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis was refractory tennis elbow;
2. Standard extracapsular method was used for surgery.

Exclusion Criteria:

1. Patient had past history of joint infection, joint tuberculosis, or osteomyelitis, or the upper limb had undergone surgery within the past 6 months;
2. Diagnosis was combined with severe heart, brain, kidney, or another organ dysfunction;
3. Case was complicated with other serious elbow joint diseases or injuries;
4. Patient did not sign the informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the quantitative data of 43 patients (14 men and 29 women) were reviewed. The minimum age was 35 years, and the maximum age was 55 years old, with an average of 44.4 years.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score | 12 months
  Use Mayo Elbow Performance Score（MEPS） to evaluate the functional recovery of patients who received extracapsular arthroscopic treatment. MEPS ranges from 0 to 100, higher scores mean a better outcome.
Visual Analog Scale | 12 months
  Use Visual Analog Scale(VAS) to evaluate the pain recovery of patients who received extracapsular arthroscopic treatment. VAS ranges from 0 to 10, higher scores mean a worse outcome.
Disability of Arm, Shoulder and Hand score | 12 months
  Use Disability of Arm, Shoulder and Hand(DASH) score to evaluate the functional and pain recovery of patients who received extracapsular arthroscopic treatment. DASH ranges from 0 to 100, higher scores mean a worse outcome.
Activity of Daily Life recovery time | 12 months
  Use Activity of Daily Life recovery time to evaluate the functional recovery of patients who received extracapsular arthroscopic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No